CLINICAL TRIAL: NCT02027584
Title: Supply of Term and Preterm Neonates With Choline, Lipids and Vitamines
Brief Title: Observational Study of Choline, Its Metabolites, and Phospholipids in Preterm Infants
Acronym: NEO-CHOLIN
Status: Completed | Type: Observational
Sponsor: University Hospital Tuebingen (Other)
Collaborators: Universität Tübingen (Other)
Responsible Party: Sponsor
Other Study IDs: NEO-CHOLIN
Record Dates: First submitted 2013-12-20; First posted 2014-01-06 (Estimated); Last update posted 2014-01-06 (Estimated); Status verified 2013-12

CONDITIONS: Prematurity
Keywords: infant, premature; infant, newborn; choline
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- parturient: mother who had given birth within 48 hours of clinically indicated blood sampling
  Interventions: Other: collection of remnant of clinically indicated blood sample
- healthy, non-pregnant, female volunteers: healthy, non-pregnant, female volunteers
  Interventions: Other: collection of remnant of clinically indicated blood sample
- preterm infant: gestational age at birth < 37 weeks
  Interventions: Other: collection of remnant of clinically indicated blood sample
- term infant: gestational age at birth >36 weeks
  Interventions: Other: collection of remnant of clinically indicated blood sample

INTERVENTIONS:
Other: collection of remnant of clinically indicated blood sample — collection of remnant of clinically indicated blood sample

SUMMARY:
To study concentrations of choline, its metabolites, and phospholipids in cord blood and remnants of clinically indicated blood samples

DETAILED DESCRIPTION:
To collect cord plasma in preterm and term infants. To collect remnants of clinically indicated blood samples in parturients and hospitalized preterm infants during neonatal intensive care.

To determine concentrations of choline, its metabolites, and phospholipids by mass spectrometry.

To compare cord plasma concentrations with postnatal plasma concentrations.

ELIGIBILITY:
Inclusion Criteria:

* meeting criteria of the 4 cohorts

Exclusion Criteria:

* none pre-defined

Max Age: 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: term and preterm neonates, parturients, non-pregnant females
Sampling Method: Non-Probability Sample
Enrollment: 414 (Actual)
Dates: Start 2008-11; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Concentration of choline in plasma | at times when a clinically indicated blood sample is taken before discharge home from the initial neonatal hospitalization (at a postnatal age of up to 4-5 months at the most in very preterm infants)

SECONDARY OUTCOMES:
concentrations of choline metabolites | at times when a clinically indicated blood sample is taken before discharge home from the initial neonatal hospitalization (at a postnatal age of up to 4-5 months at the most in very preterm infants)
Concentrations of molecular species of phosphatidylcholine and phosphatidylethanolamine | at times when a clinically indicated blood sample is taken before discharge home from the initial neonatal hospitalization (at a postnatal age of up to 4-5 months at the most in very preterm infants)

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang Bernhard, MD, PhD, Principal Investigator — University Hospital Tuebingen
Locations (1):
- University Hospital Tuebingen, Tübingen, Germany

REFERENCES:
- [Background] Bernhard W, Full A, Arand J, Maas C, Poets CF, Franz AR. Choline supply of preterm infants: assessment of dietary intake and pathophysiological considerations. Eur J Nutr. 2013 Apr;52(3):1269-78. doi: 10.1007/s00394-012-0438-x. Epub 2012 Sep 9. PMID 22961562
- [Derived] Bernhard W, Raith M, Kunze R, Koch V, Heni M, Maas C, Abele H, Poets CF, Franz AR. Choline concentrations are lower in postnatal plasma of preterm infants than in cord plasma. Eur J Nutr. 2015 Aug;54(5):733-41. doi: 10.1007/s00394-014-0751-7. Epub 2014 Aug 23. PMID 25148882